CLINICAL TRIAL: NCT01609712
Title: Osteoporotic Vertebral Compression Fractures: Can Kyphoplasty Improve Lung Function? A Prospective Evaluation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Robert Pflugmacher, PD Dr. med., University Hospital, Bonn
Other Study IDs: B-O-P-LF-01; B-O-P-LF-02 (Other: UKB Bonn, Orthopädie und Unfallchirurgie, PD Dr. Robert Pflugmacher)
Record Dates: First submitted 2012-05-29; First posted 2012-06-01 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Osteoporotic Vertebral Compression Fractures; Lung Function
Keywords: Improvement of lung function (FEV1, PEF); Visual Analog Scale; Oswestry Disability Index; Radiographs pre and post Op

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient with vertebral compression fracture: RF kyphoplasty is standard of care in our hospital for patients with osteoporortic compression fractures. We are intersetd, if it also can improve the lung function.
  Interventions: Procedure: Radiofrequency Kyphoplasty

INTERVENTIONS:
Procedure: Radiofrequency Kyphoplasty — Radiofrequency kyphoplasty is a new form of surgical treatment. It injects an ultrahigh viscosity cement into the fractured vertebral body, using radiofrequency to achieve the proper consistency of the cement. This ultrahigh viscosity cement is designed to first restore proper height and alignment to the fractured vertebra and then to stabilize the fracture, thereby preventing further intravertebral motion and reducing pain.
  The RF-Kyphoplasty is standard of care in our hospital. It is FDA and CE approved.
  Other Names: RF-Kyphoplasty

SUMMARY:
Patients with vertebral fractures often have problems to straighten and as a consequence of impaired lung ventilation that leads to a impaired lung function. Furthermore, it comes to the sintering of the vertebra and a so-called hunchback. This also contributes to the poorer expansion of the lung. Pain is also caused by respiratory excursions of the chest which hinder the patients to use their entire lung volume.

Kyphoplasty is designed to counter all these consequences of vertebral fractures by bringing stability to the fracture.

In order to prove the thesis the results of lung function test (FEV1, PEF) are assessed.

ELIGIBILITY:
Inclusion Criteria:

* over 50 years
* VAS over 49, ODI over 29
* radiographic evidence of A 1.1, 1.2, 1.3 fractures
* patients mentally capable to sign informed consent

Exclusion Criteria:

* high-energy trauma
* known tumor involvement
* osteonecrotic fractures
* burst fractures or pedicle fractures
* previous surgical treatment for a vertebral body compression fracture
* patient has paget's disease
* BMI > 35
* uncontrolled diabetes HbAc1c > 7%
* severe cardiopulmonary disease
* Myelopathy
* long-time steroid therapy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with osteoporotic compression fractures, mostly elderly females
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-05

CONTACTS AND LOCATIONS:
Overall Officials: Robert Pflugmacher, M.D., Principal Investigator — Orthopädie und Unfallchirurgie, Universitätsklinkum Bonn
Locations (1):
- Orthopädie und Unfallchirurgie Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia, Germany